CLINICAL TRIAL: NCT06688422
Title: Incentive Spirometry for Respiratory Enhancement Pilot Clinical Trial in Lung Cancer Patients Undergoing Concurrent Chemotherapy and Radiation Therapy
Brief Title: Incentive Spirometry to Improve Outcomes in Lung Cancer Patients Undergoing Concurrent Chemotherapy and Radiation Therapy
Acronym: INSPIRE-CRT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cooper Health System (Other)
Collaborators: The Cooper Foundation (Unknown)
Responsible Party: Principal Investigator, Veli Bakalov, Assistant Professor of Medicine, Cooper Medical School of Rowan University, The Cooper Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-135
Record Dates: First submitted 2024-11-09; First posted 2024-11-14 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancer; Pneumonitis; Radiation-Induced Lung Injury; Immunotherapy-Induced Pneumonitis; Non-Small-Cell Lung Cancer (NSCLC)
Keywords: Incentive Spirometry; Chemotherapy; Radiation Therapy; Quality of Life (QoL); Respiratory Complications; Advanced Lung Cancer; Concurrent Chemoradiotherapy; Pulmonary Toxicity; Immunotherapy Maintenance; Lung Function
MeSH Terms: conditions — Lung Neoplasms; Pneumonia; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Intervention Arm (Experimental): The study will have one intervention group of patients using incentive spirometry in addition to standard of care treatment, including chemo/radiation and immunotherapy maintenance. For research purposes, patients will be asked to use incentive spirometry. Patients will use the incentive spirometer 10 times (10 breaths) every hour they are awake. Patients will be asked to start using the incentive spirometer as soon as they are enrolled in the study. Patients will be asked to continue to use incentive spirometry daily, including the duration of chemoradiation and up to three months post-treatment. Patients will be asked to to complete QoL assessments.
  Interventions: Device: incentive spirometry

INTERVENTIONS:
Device: incentive spirometry — The study will have one intervention group of patients using incentive spirometry in addition to standard of care treatment, including chemo/radiation and immunotherapy maintenance. Patients will use the incentive spirometer 10 times (10 breaths) every hour they are awake. Patients will be asked to start using the incentive spirometer as soon as they are enrolled in the study. Patients will be asked to continue to use incentive spirometry daily, including the duration of chemoradiation and up to three months post-treatment.

SUMMARY:
The goal of this clinical trial is to learn if using an incentive spirometer can reduce lung problems in people with advanced lung cancer who are receiving chemotherapy and radiation therapy. The main questions the study aims to answer are:

Does using an incentive spirometer lower the chances of developing lung inflammation (pneumonitis)? Does it improve overall survival and quality of life?

Participants will:

Use an incentive spirometer, a device that helps with deep breathing, 10 times every hour while awake.

Continue using the spirometer daily during treatment and for up to three months after treatment.

Complete quality of life assessments at the start of the study and at 3, 6, and 12 months.

Researchers will compare the results to see if the incentive spirometer helps reduce lung problems and improves participants' well-being during and after their cancer treatment.

DETAILED DESCRIPTION:
The INSPIRE-LUNG-CRT trial is a prospective, pilot study investigating the efficacy of incentive spirometry on the incidence and severity of pneumonitis in lung cancer patients undergoing concurrent chemotherapy and radiation therapy with immunotherapy maintenance. Despite advancements in treatment modalities, pulmonary complications remain a significant challenge, often leading to diminished functional capacity and quality of life. The trial aims to establish incentive spirometry as a non-pharmacological intervention to reduce these complications, thereby improving clinical outcomes and patient well-being. Lung cancer treatments are frequently associated with pulmonary toxicities, such as radiation-induced pneumonitis and fibrosis, immunotherapy induced pneumonitis, significantly impacting patient outcomes. Incentive spirometry, a device that encourages deep breathing and lung expansion, has shown promise in postoperative settings but is underutilized in oncology.

The pilot, prospective trial will enroll 100 patients diagnosed with advanced, unresectable non-small-cell lung cancer, candidates will receive concurrent chemotherapy and radiation therapy. Inclusion criteria includes a confirmed diagnosis of advanced non-small-cell lung cancer, good performance status (ECOG 0-1), and eligibility for concurrent chemotherapy and radiation. Exclusion criteria includes previous lung or thoracic surgery, enrollment in another pulmonary intervention trial, home oxygen usage prior to enrollment, radiological evidence of pleural effusion, pneumothorax, bullous emphysema, or pneumonitis, active respiratory tract infection, uncontrolled nausea and vomiting, prior exposure to certain drugs, and inability to give informed consent.

The primary endpoint is to determine the impact of incentive spirometry on the incidence and severity of pneumonitis. Secondary endpoints include evaluating the impact on overall survival and patients' quality of life using the EORTC QLQ-C30 questionnaire. Patients will use the incentive spirometer 10 times (10 breaths) every hour while awake, starting as soon as they are enrolled in the study. The use will continue daily during chemoradiation and up to three months post-treatment. The study duration for each subject is approximately six months, including the use of incentive spirometry during the concurrent chemoRT phase (6-8 weeks) and continued use for up to three months post-treatment.

Inclusion Criteria:

* Confirmed diagnosis of advanced non-small-cell lung cancer
* Performance status (ECOG 0-1)
* Eligible for concurrent chemotherapy and radiation
* 18 years or older.

Exclusion Criteria:

* Previous lung or thoracic surgery
* Enrollment in another pulmonary intervention trial
* Home oxygen usage prior to enrolment
* Radiological evidence of pleural effusion, pneumothorax, bullous emphysema, or pneumonitis on staging imaging
* Presence of active respiratory tract infection
* Uncontrolled nausea and vomiting
* Prior exposure to drugs such as amiodarone, bleomycin, or immunotherapy
* Inability or unwillingness of individual to give written informed consent

Interventions The study will have one intervention group of patients using incentive spirometry in addition to standard of care treatment, including chemo/radiation and immunotherapy maintenance. Patients will undergo procedures for diagnostic and treatment purposes. Standard procedures for lung cancer patients includes, but is not limited to, routine diagnostic tests such as imaging (CT scans, PET scans, MRI scan), blood tests, and pulmonary function tests (PFTs), diagnostic biopsies. For research purposes, patients will be asked to use incentive spirometry. Patients will use the incentive spirometer 10 times (10 breaths) every hour they are awake. Patients will be asked to start using the incentive spirometer as soon as they are enrolled in the study. Patients will be asked to continue to use incentive spirometry daily, including the duration of chemoradiation and up to three months post-treatment. Patients will be asked to monitoring adherence to the spirometry regimen through patient logs and periodic check-ins.

Duration of Participation. The study duration for each subject is approximately 12 months, including: Use of incentive spirometry during the concurrent chemoRT phase (approximately 6-8 weeks). Continued use of the spirometer for up to three months post-treatment. Quality of life assessments and pulmonary function tests at 3-, 6- and 12 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of advanced non-small-cell lung cancer
* Performance status (ECOG 0-1)
* Eligible for concurrent chemotherapy and radiation
* 18 years or older

Exclusion Criteria:

* Previous lung or thoracic surgery
* Enrollment in another pulmonary intervention trial
* Home oxygen usage prior to enrolment
* Radiological evidence of pleural effusion, pneumothorax, bullous emphysema, - or pneumonitis on staging imaging
* Presence of active respiratory tract infection
* Uncontrolled nausea and vomiting
* Prior exposure to drugs such as amiodarone, bleomycin, or immunotherapy
* Inability or unwillingness of individual to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Pneumonitis | 12 months
  Primary Endpoint: To determine the impact of incentive spirometry on the incidence of pneumonitis.
  Assessment Method: Number of participants diagnosed with pneumonitis, assessed using CT scan and clinical diagnostic criteria

SECONDARY OUTCOMES:
Number of Patients with Severe Pneumonitis | 12 months
  Secondary Endpoint: To determine the impact of incentive spirometry on the severity of pneumonitis.
  Assessment Method: number of patients diagnosed with severe pneumonitis, evaluated using a standardized CTCAE grading (Common Terminology Criteria for Adverse Events)

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson Cancer Center at Cooper, Camden, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data (IPD) due to privacy concerns and the need to protect the confidentiality of participants. Additionally, the data collected during this study includes sensitive health information that could potentially identify participants, even when de-identified. Given the nature of the data and ethical considerations, we have decided not to make IPD available to other researchers.

REFERENCES:
- [Background] Vansteenkiste JF, Naidoo J, Faivre-Finn C, Ozguroglu M, Villegas A, Daniel D, Murakami S, Hui R, Lee KH, Cho BC, Kubota K, Broadhurst H, Wadsworth C, Newton M, Thiyagarajah P, Antonia SJ. Symptomatic Pneumonitis With Durvalumab After Concurrent Chemoradiotherapy in Unresectable Stage III NSCLC. JTO Clin Res Rep. 2024 Jan 18;5(3):100638. doi: 10.1016/j.jtocrr.2024.100638. eCollection 2024 Mar. PMID 38455595
- [Background] Zhong L, Altan M, Shannon VR, Sheshadri A. Immune-Related Adverse Events: Pneumonitis. Adv Exp Med Biol. 2020;1244:255-269. doi: 10.1007/978-3-030-41008-7_13. PMID 32301020